CLINICAL TRIAL: NCT05381376
Title: Multicentre Prospective Clinical Database for the Construction of Predictive Models on Risk of Intrauterine Adhesion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hua Duan (Other)
Responsible Party: Sponsor-Investigator, Hua Duan, Director of Minimally Invasive Gynecologic Center, Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing Obstetrics and Gynecology Hospital
Organization: Beijing Obstetrics and Gynecology Hospital (Other)
Other Study IDs: IUADB
Record Dates: First submitted 2022-05-08; First posted 2022-05-19 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Database for Intrauterine Adhesion; Risk Factors for Intrauterine Adhesion; Risk Stratification and Prognostic Assessment; Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia | interventions — Hysteroscopy; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hysteroscopy — Hysteroscopy for CSGE, AFS, and endometrial receptivity assessment
Diagnostic Test: Ultrasonography — Ultrasonography for Uterus size and endometrial thickness

SUMMARY:
1. To establish a follow-up database for uterine adhesions and a library of biological specimens for Intrauterine Adhesion. 2. using epidemiological surveys and biological analyses to screen risk factors for the development and prognosis of Intrauterine Adhesion. 3. Predictive models based on clinical and biochemical indicators, specimen testing and hysteroscopic images are also combined with statistical analysis and machine learning algorithms to enable patients' risk stratification and prognostic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnostic hysteroscopy confirmed adhesions combined with infertility or recurrent pregnancy loss (early pregnancy loss >2)
* Desiring to conceive
* Ages between 20-45 years;
* Patients without gynecological endocrine disorders (e.g. PCOS) and AMH>1ng/ml;
* Signing informed consent.

Exclusion Criteria:

* Hysteroscopy contraindications;
* Hormone therapy contraindications;
* Pregnancy contraindications;
* History of malignant pelvic tumor and radiotherapy;
* Severe hepatic or renal dysfunction;
* Complicated with hematological disorders (eg.platelet dysfunction, severe anemia, blood-borne infections);
* Male factor infertility(eg.seminal abnormalities).

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Taking α=0.05 and β=0.1, the overall time incidence (pregnancy rate) was taken as the lowest value of P=0.25, the risk factor (uterine adhesion fraction) coefficient was -0.18, and the decision coefficient for the risk factor (uterine adhesion fraction) was 0.8. The PASS software calculated 1622, taking into account the shedding factor (20%) and the randomization requirement of n=2028, based on each center's outpatient volume, the total number of cases to be included in this study database is at least 2200.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Rate of pregnancy | 2 years

SECONDARY OUTCOMES:
Recurrence rate of IUA | 3 month
  Recurrence rate of Intrauterine Adhesion
Menstrual blood volume | 3 month
CSGE | 3 month
  CSGE (Chinese Society of Gynaecological Endoscopy score), scale 0-28, higher scores mean a worse outcome
AFS | 3 month
  AFS(American Fertility Association score), scale 1-12, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Yishaofu Hospital, Hangzhou, Zhejiang
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing